CLINICAL TRIAL: NCT06547385
Title: ONO-4578 Phase I Study An Open-label, Uncontrolled Study of First-line Combination Therapy of ONO-4578 and ONO-4538 With Standard Therapy XELOX Plus Bevacizumab or FOLFOX Plus Bevacizumab in Patients With Unresectable, Advanced or Recurrent Colorectal Cancer
Brief Title: Study of ONO-4578 and XELOX/FOLFOX Plus Bevacizumab in Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4578-02
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nivolumab; Capecitabine; Oxaliplatin; Fluorouracil; Leucovorin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONO-4578+ONO-4538+XELOX plus bevacizumab (Experimental)
  Interventions: Drug: ONO-4578; Drug: ONO-4538; Drug: Capecitabine; Drug: Oxaliplatin; Drug: Bevacizumab
- ONO-4578+ONO-4538+FOLFOX plus bevacizumab (Experimental)
  Interventions: Drug: ONO-4578; Drug: ONO-4538; Drug: Oxaliplatin; Drug: Fluorouracil; Drug: Calcium Levofolinate Hydrateb; Drug: Bevacizumab

INTERVENTIONS:
Drug: ONO-4578 — Specified dose on specified days
Drug: ONO-4538 — Specified dose on specified days
  Other Names: Nivolumab
Drug: Capecitabine — Specified dose on specified days
  Other Names: XELODA
  Arms: ONO-4578+ONO-4538+XELOX plus bevacizumab
Drug: Oxaliplatin — Specified dose on specified days
  Other Names: ELPLAT
Drug: Fluorouracil — Specified dose on specified days
  Other Names: 5-FU
  Arms: ONO-4578+ONO-4538+FOLFOX plus bevacizumab
Drug: Calcium Levofolinate Hydrateb — Specified dose on specified days
  Other Names: ISOVORIN
  Arms: ONO-4578+ONO-4538+FOLFOX plus bevacizumab
Drug: Bevacizumab — Specified dose on specified days
  Other Names: AVASTIN

SUMMARY:
To evaluate the tolerability and safety of combination of ONO-4578 and ONO-4538 and the standard of care XELOX + bevacizumab or the safety of combination of ONO-4578 and ONO-4538 and the standard of care FOLFOX + bevacizumab as first-line therapy in patients with unresectable, advanced, or recurrent colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable colorectal cancer
* Life expectancy of at least 3 months
* Patients with ECOG performance status 0 or 1

Exclusion Criteria:

* Patients with severe complication
* Patients are unable to swallow oral medications

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of AEs and SAEs | up to 3years
Incidence and severity of clinical laboratory abnormalities | up to 3years
12-lead electrocardiography (Heart rate) | up to 3years
12-lead electrocardiography (PR interval) | up to 3years
12-lead electrocardiography (RR interval) | up to 3years
12-lead electrocardiography (QRS width) | up to 3years
12-lead electrocardiography (QT interval) | up to 3years
Chest X-ray test | up to 3years
ECOG performance status | up to 3years

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 3years
Disease control rate (DCR) | up to 3years
Overall survival (OS) | up to 3years
Progression-free survival (PFS) | up to 3years
Duration of response (DOR) | up to 3years
Time to response (TTR) | up to 3years
Best oveall response (BOR) | up to 3years
Percentage of change in the sum of tumor diameters of target lesions | up to 3years
Maximum percent change in the sum diameters of the target lesions | up to 3years
Time course of tumor markers | up to 3years
Plasma ONO-4578 concentration | up to 3years
Serum ONO-4538 concentration | up to 3years
Anti-ONO-4538 antibody | up to 3years

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (9):
- Japan (9):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Kobe City Hospital Organization Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Saitama Cancer Center, Ina, Kitaadati-gun, Saitama
  - NHO Osaka National Hospital, Osaka, Osaka
  - Osaka General Medical Center, Osaka, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki-shi, Osaka
  - Saitama Medical University International Medical Center, Hidaka-shi, Saitama
  - Cancer Institute Hospital of JFCR, Koto-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No